CLINICAL TRIAL: NCT06833125
Title: The Prophylactic Effect of Garlic Tablets to Prevent Nosocomial Infections in Intensive Care Unit Patients.
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0108752
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-02

CONDITIONS: Nosocomial Infection
Keywords: nosocmial infection; prophylaxis; garlic
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: It is a randomized non blinded controlled trial. Eligible patients will be randomly divided into two groups: An intervention group which will receive garlic tablets (Tomex plus 300 mg) two tablets twice daily for 6 days just after ICU admission and a control group which will not receive the garlic tablets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The intervention group (Experimental): The patients in the intervention group which will receive garlic tablets (Tomex plus 300 mg) two tablets twice daily for 6 days just after ICU admission
  Interventions: Drug: Garlic powder standardized to allicin
- The control group (No Intervention): The patients in the control group which will not receive the garlic tablets.

INTERVENTIONS:
Drug: Garlic powder standardized to allicin — The intervention is the administration of garlic tablets (Tomex plus 300 mg) two tablets twice daily (which contains 5.4 mg allicin the active ingredient with anibacterial effect) for 6 days just after ICU admission
  Arms: The intervention group

SUMMARY:
The goal of this clinical trial is to learn if garlic tablets works to prevent nosocomial infections in hospitalized patients in ICU. The main questions it aims to answer are:

Does garlic tablets administration lower the occurence of nosocomial infections in hospitalized patients in ICU?

ELIGIBILITY:
Inclusion Criteria:

* All patients aged from 18 to 65 years old admitted to intensive care units without any type of infection.

Exclusion Criteria:

1. Patients with signs /symptoms of infection.
2. Patients with human immunodeficiency virus, malignancy and patients with a history of recent immunosuppressants or corticosteroids administration.
3. Patients with bleeding disorders or abnormal coagulation profile
4. Patients who will planned for surgery within 2 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of central line-associated bloodstream infections, catheter- associated urinary tract infections, surgical site infections and ventilator- associated pneumonia in the two groups (by cultures results). | one year

SECONDARY OUTCOMES:
Values of Blood white cell count, body temperature and C-reactive protein of the patient in the two groups . | one year
  The Mean of Blood white cell count (number per micro liter) , body temperature ( by the degree Celsius) and C-reactive protein (milligrams per liter ) of the patients in the two groups will be calculated.
Values of Blood white cell count, body temperature and C-reactive protein of the patient in the two groups . | one year
  The Mean of Blood white cell count, body temperature and C-reactive protein of the patient in the two groups will be calculated.

OTHER OUTCOMES:
Antibiotics consumption as total number of vials per each antibiotic in the two groups. | one year
Lenghth of stay of patients in ICU (by average number of days) in the two groups | one year
Mortality rate of patients in the two groups | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospital, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided